CLINICAL TRIAL: NCT02262793
Title: Relative Bioavailability of Telmisartan in Micardis® and of Dipyridamole in Aggrenox® After Co-administration Compared to the Bioavailability of Telmisartan Respectively of Dipyridamole After Oral Administration of 80 mg Telmisartan Respectively of 25 mg ASA/200 mg Extended-release Dipyridamole Alone. An Open-label, Randomised, Single-dose, Four-way Crossover Study in 24 Healthy Female and Male Subjects
Brief Title: Relative Bioavailability of Telmisartan and Dipyridamole After Co-administration Compared to the Bioavailability of Telmisartan or Dipyridamole Alone in Healthy Female and Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.458
Record Dates: First submitted 2014-10-10; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan

ARMS (4):
- telmisartan and ASA/ER-DP (concomitant) (Experimental)
  Interventions: Drug: telmisartan; Drug: ASA/ER-DP
- ASA/ER-DP alone (Active Comparator)
  Interventions: Drug: ASA/ER-DP
- telmisartan and ASA/ER-DP (consecutively) (Experimental)
  Interventions: Drug: telmisartan; Drug: ASA/ER-DP
- telmisartan (Active Comparator)
  Interventions: Drug: telmisartan

INTERVENTIONS:
Drug: telmisartan
  Arms: telmisartan; telmisartan and ASA/ER-DP (concomitant); telmisartan and ASA/ER-DP (consecutively)
Drug: ASA/ER-DP
  Arms: ASA/ER-DP alone; telmisartan and ASA/ER-DP (concomitant); telmisartan and ASA/ER-DP (consecutively)

SUMMARY:
To investigate the relative bioavailability of telmisartan respectively of dipyridamole after concomitant administration of 80 mg telmisartan in Micardis® and 25 mg acetylsalicylic acid (ASA)/200 mg extended release (ER) dipyridamole (DP) in Aggrenox® (Test 1) relative to ER-DP in Aggrenox® alone (Reference 1), respectively relative to telmisartan in Micardis® alone (Reference 2).

To investigate the relative bioavailability of dipyridamole respectively of telmisartan administered as 25 mg ASA/200 mg ER-DP 30 minutes after intake of 80 mg telmisartan (Test 2) relative to dipyridamole in Aggrenox® alone (Reference 1), respectively relative to telmisartan in Micardis® alone (Reference 2).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy females and males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, HR), 12-lead ECG, clinical laboratory tests
   * No finding deviating from normal and of clinical relevance
   * No evidence of a clinically relevant concomitant disease
2. Age ≥21 and Age ≤65 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts.
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
7. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
8. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
9. Participation in another trial with an investigational drug within two months prior to administration or during the trial
10. Smoker (more than 10 cigarettes/day or 3 cigars/day or 3 pipes/day)
11. Inability to refrain from smoking on trial days
12. Alcohol abuse (more than 60 g/day)
13. Drug abuse
14. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
15. Excessive physical activities (within one week prior to administration or during the trial)
16. Any laboratory value outside the reference range that is of clinical relevance
17. Inability to comply with dietary regimen of study centre
18. History of hereditary fructose intolerance
19. History of any familial bleeding disorder
20. Veins unsuited for i.v. puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture, etc.)
21. Inability to comply with the investigators instructions

    For female subjects:
22. Pregnancy
23. Positive pregnancy test
24. No adequate contraception e.g. oral contraceptives, sterilization, intrauterine device (IUD)
25. Inability to maintain this adequate contraception during the whole study period
26. Lactation period

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-05; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration time curve in plasma from 0 extrapolated to infinity) | up to 72 hours following drug administration
Cmax (maximum concentration in plasma) | up to 72 hours following drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours following drug administration
AUCt1-t2 (Area under the concentration time curve in plasma over the time interval t1 to t2) | up to 72 hours following drug administration
tmax (time from dosing to the maximum concentration of the analytes in plasma) | up to 72 hours following drug administration
λz (terminal rate constant in plasma) | up to 72 hours following drug administration
t1/2 (terminal half-life of the analytes in plasma) | up to 72 hours following drug administration
MRTpo (mean residence time of the analyte in the body after p.o. administration) | up to 72 hours following drug administration
CL/F (apparent clearance of the analytes in the plasma after extravascular administration) | up to 72 hours following drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours following drug administration
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with clinically significant findings in vital signs | up to 8 days after last drug administration
  blood pressure, heart rate
Number of subjects with clinically significant findings in 12 lead ECG | up to 8 days after last drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 8 days after last drug administration
Assessment of tolerability by the investigator on a 4-point scale | up to 8 days after last drug administration